CLINICAL TRIAL: NCT01165970
Title: Vergleichende, Randomisierte, Kontrollierte Und Doppelblinde In-situ-Studie Zur Wirkung Von Speichelersatzmitteln Auf Schmelz Und Dentin
Brief Title: Effect of Saliva Substitutes on Dental Hard Tissues in Situ
Acronym: T-01
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Peter Tschoppe, Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: T-01/2008-005451-23; 2008-005451-23 (EudraCT Number)
Record Dates: First submitted 2010-06-30; First posted 2010-07-20 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Hyposalivation
Keywords: enamel; dentin; saliva substitute; demineralization; remineralization
MeSH Terms: conditions — Xerostomia | interventions — Glandosane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glandosane (Active Comparator): After in situ exposition the enamel and dentin samples will demineralize with Glandosane.
  Interventions: Drug: Glandosane
- Saliva natura (Experimental): After in situ exposition the enamel and dentin samples will remineralize with Saliva natura
  Interventions: Device: Saliva natura

INTERVENTIONS:
Drug: Glandosane — according to the german law the sued saliva substitute is a drug (Glandosane) whereas Saliva natura is a medical product
  Other Names: Glandosane, Cell Pharm, Germany
  Arms: Glandosane
Device: Saliva natura — Saliva substitute without restriction to be used
  Other Names: Saliva natura, Medac, Germany
  Arms: Saliva natura

SUMMARY:
Symptomatic hyposalivation is associated not only with Sjögren's syndrome or salivary gland hypofunction in elderly patients, but also with medications containing antimuscarinic drugs, chemo radiotherapy for head and neck carcinomas, and psychiatric disorders (Atkinson & Ava, 1994, Kielbassa et al., 2006).

Human saliva possesses important physiological functions in protecting and moistening the oral hard and soft tissues (Piotrowski et al., 1992, ). Consequently, decreasing salivation causes oral dysfunction and promotes severe oral side effects (reduced antibacterial function, lack of remineralisation, reduced buffer capacity) (Tschoppe et al., 2010a). These have been identified as being responsible for the rapid destruction of the dentition (Willich et al., 1988). Saliva substitutes are frequently applied for relieving the symptoms in patients suffering from hyposalivation (Hahnel et al., 2009, Nieuw Amerongen & Veerman, 2003, Vissink et al., 2004). Besides the moistening and lubrication of the oral mucosa, these products should also protect dental hard tissues. However, in vitro studies revealed that some marketed products have only a neutral or even a demineralising potential on enamel as well as on dentin (Kielbassa et al., 2001, Meyer-Lueckel et al., 2002, Smith et al., 2001, Tschoppe et al., 2009). Inorganic ions such as calcium, phosphates, and fluorides have been added to saliva substitutes in order to enhance their remineralising property or minimize their demineralising potential (Tschoppe et al., 2009). Furthermore, as most patients suffering from hyposalivation are elderly people, recessions and subsequently exposed dentin surfaces are very common. Since dentin is not as acid resistant as enamel, an earlier and more severe demineralisation can be expected (Saunders & Meyerowitz, 2005).

Therefore, the current in situ study was performed to assess the effects of a demineralising and a remineralising saliva substitutes on the mineralisation of dental hard tissues. It was hypothesized that storage in Glandosane(cell pharm, Hannover, Germany) would not result in pronounced mineral loss of dentin specimens, and that storage in Saliva natura would not result in enhanced remineralisation when combined with a remineralising artificial saliva (Saliva natura supersaturated with respect to relevant calcium phosphates; medac, Hamburg, Germany) (H0). These null hypotheses were tested against the alternative hypothesis of a difference.

DETAILED DESCRIPTION:
see application for the German Federal Institute for Drugs and Medical Devices at Eudra-CT

ELIGIBILITY:
Inclusion Criteria:

* stimulated salivary flow rate < 0.5 ml/min
* partial denture upper or lower jaw
* radiationtherapy in the head and neck area
* patient age above 18 years
* Signed informed consent (AMG §40 (1) 3b)

Exclusion Criteria:

* stimulated salivary flow rate > 0.5 ml/min
* missing partial denture upper or lower jaw
* missing Radiationtherapy in the head and neck area
* paraben allergy
* not signed informed consent (AMG §40 (1) 3b)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Mineral loss and lesion depth of specimens | 15 weeks
  Evaluation of the mineral loss/lesion depth of the enamel and dentin specimens after in situ exposition evaluated with transversal microradiography. The Unit is the mineral oss as well as lesion depth.

SECONDARY OUTCOMES:
general and oral well being | 15 weeks
  Evaluation of the general and oral well being before and after therapy by questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tschoppe, Dr, Principal Investigator — Department of Operative Dentistry and Periodontology, School of Dental Medicine, CharitéCentrum 3, Charité - Universitätsmedizin Berlin
Locations (2):
- Germany (2):
  - Charite, Berlin, Germany, Berlin, State of Berlin
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin

REFERENCES:
- [Derived] Tschoppe P, Wolf O, Eichhorn M, Martus P, Kielbassa AM. Design of a randomized controlled double-blind crossover clinical trial to assess the effects of saliva substitutes on bovine enamel and dentin in situ. BMC Oral Health. 2011 Apr 9;11:13. doi: 10.1186/1472-6831-11-13. PMID 21477333
- See also: please check the science subsite — http://kons-paro.charite.de
- See also: Short review on the main problems in this patient population: Etiologic factors of hyposalivation and consequences for oral health. Quintessence Int. 2010 Apr;41(4):321-33. Review. — http://www.ncbi.nlm.nih.gov/pubmed/20305867